CLINICAL TRIAL: NCT06827158
Title: Validity and Reliability Study of the Turkish Version of the Manual Dexterity Questionnaire for Parkinson's Patients-24 (DextQ-24)
Brief Title: Validity and Reliability of the Turkish Version of the Manual Dexterity Questionnaire
Status: Enrolling by invitation | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Gulhan Yilmaz Gokmen, Assos. Prof., Bandırma Onyedi Eylül University
Other Study IDs: 2024-186
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease; Validation Studies; Dexterity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: validity and reliability of the Turkish version of the Dexterity Questionnaire 24 (DextQ-24 — Permission for the Turkish translation and validation of the DextQ-24 questionnaire was obtained from its developer, Tim Vanbellingen. The original English version will be translated into Turkish by two independent translators and then back into English by two native English speakers. After review, the finalized version will be used in the study.
  Patients diagnosed with Parkinson's disease (aged 40-80) will complete consent and demographic forms. The Mini-Mental State Examination (MMSE) will exclude those scoring ≤24. Disease staging will follow the Hoehn and Yahr Scale (stages I-IV included). The MDS-UPDRS (sections II and III) will assess disease severity, while the Nine-Hole Peg Test and Hand Dexterity Scale-36 will evaluate hand function. Participants will complete the Turkish DextQ-24, with 30 randomly selected patients retaking it after two weeks for reliability testing. Data collection per participant will take approximately 30 minutes.

SUMMARY:
El fonksiyonunun bozulması, özellikle ince motor becerileri gerektiren aktivitelerde önemli zorluklara yol açar. Parkinson hastalığı teşhisi konan bireylerin yaklaşık %90'ı, gömleği düğmelemek, ayakkabı bağcıklarını bağlamak veya bozuk paralarla uğraşmak gibi elli görevleri yerine getirmekte zorluk çeker. Ambülasyon zorlukları ve bilişsel bozukluğun ardından, el fonksiyonundaki eksiklikler Parkinson hastalığı olan bireylerde yaşam kalitesini olumsuz etkileyen üçüncü en önemli faktörü temsil eder. El Beri Anketi (DextQ-24), Parkinson hastalığı olan bireylerde, özellikle günlük aktiviteler bağlamında el fonksiyonunu değerlendirmek için geçerli ve güvenilir bir araç olarak tanımlanmıştır. Bununla birlikte, mevcut literatürün gözden geçirilmesi ve anketin orijinal geliştiricisi ile doğrudan iletişim, bir Türkçe çevirinin henüz doğrulanmadığını veya güvenilirlik açısından test edilmediğini göstermektedir.

Bu çalışmanın amacı, Parkinson hastalığı olan bireylerde el fonksiyonunun değerlendirilmesi için El Beceri Anketi'nin (DextQ-24) Türkçe versiyonunun geçerliliğini ve güvenilirliğini değerlendirmek, böylece klinik uygulamada, değerlendirmelerde ve gelecekteki araştırmalarda kullanımını kolaylaştırmaktır.

DETAILED DESCRIPTION:
Nörolojik hastalıklar sıklıkla el performansını etkileyerek fonksiyonel sakatlıklara yol açar. Bunlar arasında Parkinson hastalığı, el fonksiyonu üzerinde önemli bir etkisi olan hem motor hem de motor olmayan semptomlarla karakterize kronik, ilerleyici bir nörodejeneratif bozukluktur. Hastalık öncelikle substantia nigra'da dopaminerjik nöronların dejenerasyonu veya kaybı ile ilişkilidir ve genellikle orta yaşlı ve yaşlı bireylerde görülür ve başlangıç tipik olarak 50 ila 60 yaşları arasında meydana gelir. Dinlenme titremesi, sertlik, postural instabilite ve bradikinezi gibi motor semptomlar birincil klinik tanı kriterlerini oluşturur. Bradikinezi veya hareket yavaşlığı, yatakta dönme veya oturma pozisyonundan ayakta durma da dahil olmak üzere motor görevleri yerine getirmede zorluklara katkıda bulunur. Ek olarak, nesne manipülasyonunda bozulmalar ve el-parmak koordinasyonunda bir düşüş sıklıkla gözlenmektedir. El fonksiyonunun bozulmasının altında yatan kesin mekanizmalar belirsiz kalsa da, bradikinezi, kas güçsüzlüğü ve azalmış parmak momentumu gibi motor bozuklukların katkıda bulunan faktörler olduğuna inanılmaktadır. El fonksiyonu, Parkinson hastalığının çeşitli aşamalarında günlük ve fonksiyonel aktivitelerin yürütülmesinde çok önemli bir rol oynar.

Assessment and training of hand functions constitute a significant component of treatment approaches in the field of physiotherapy and rehabilitation. Fine and gross motor skills, as well as hand outcome measures, play a crucial role in evaluating hand functions. Various standardized tests, including the Jebsen Taylor Hand Function Test, the Nine-Hole Peg Test, the Purdue Pegboard Test, and the Minnesota Manual Dexterity Test, are commonly used for this purpose. However, assessment tools and questionnaires specifically designed to evaluate hand function in the context of daily living activities remain limited. One such measure is the Hand Skills Questionnaire-36 (HSQ-36), which has been translated into Turkish and validated for reliability. In this study, the validity and reliability of the Turkish version of the Dexterity Questionnaire 24 will be tested using the HSQ-36 and the Nine-Hole Peg Test.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study voluntarily
* A confirmed diagnosis of Parkinson's disease
* Age range between 40 and 80 years
* Disease stage classified as Hoehn & Yahr Stage I-IV
* Mini-Mental State Examination (MMSE) score >24

Exclusion Criteria:

* Presence of any neurological disease other than Parkinson's disease (e.g., multiple sclerosis, muscular disorders, stroke)
* History of any surgical procedure involving the upper extremities
* Presence of hand deformities unrelated to Parkinson's disease (e.g., rheumatoid arthritis, nerve injury, connective tissue disorders)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Dexterity Questionnaire (DextQ-24) | 5 minutes
  The questionnaire examines hand functions under five main categories: washing and grooming, dressing, eating and kitchen tasks, daily activities, and TV-CD-DVD usage. Performing a function without difficulty is scored as 1, while being unable to perform the function without external assistance is scored as 4. The total score ranges from 24 to 96. The questionnaire, whose validity and reliability have been investigated in Parkinson's patients, has been shown to be valid and reliable.
Manual Ability Measure (MAM-36) | 5 minutes
  MAM-36 is a tool developed to assess hand function in rehabilitation patients. The scale consists of 36 activities and uses a scoring system ranging from 1 to 4, where 1 indicates that the activity cannot be performed, and 4 indicates that it is performed easily (Proud et al., 2019). A Turkish validity and reliability study has been conducted for neurological patients, demonstrating excellent test-retest reliability (ICC: 0.94) and high internal consistency (Cronbach's Alpha: 0.94).
The Nine Hole Peg Test (NHPT) | 2 minute
  The Nine Hole Peg Test (NHPT) involves placing and removing nine pegs and is used to assess fine hand dexterity. The test-retest reliability was found to be ICC: 0.88 for the dominant hand and ICC: 0.91 for the non-dominant hand. It has been identified as a useful assessment tool for evaluating upper extremity function in Parkinson's patients.

SECONDARY OUTCOMES:
The Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 20 minutes
  MDS-UPDRS, developed in 1980, is widely used in clinical studies and consists of four sections. The first section assesses cognition, behavior, and mood, the second section evaluates activities of daily living, and the fourth section focuses on motor complications, all based on patient and caregiver-reported questionnaires. The third section provides an objective evaluation of the patient's motor abilities. Each item is scored between 0 and 4, with higher scores indicating greater disease severity.
  In 2001, a modified version, the MDS-UPDRS, was introduced. This version consists of 50 items: 13 questions on non-motor experiences (Section 1), 13 questions on motor experiences (Section 2), 18 items assessing motor function (Section 3), and 6 items on motor complications (Section 4). Unlike the original scale, it replaces the term "activities" with "experiences." Scoring remains on a 0 to 4 scale.
Mini-Mental State Examination (MMSE) | 10 minutes
  The Mini-Mental State Examination (MMSE) consists of five subcategories: orientation (each question 1 point, total 10 points), immediate recall (3 points), attention and calculation (5 points), recall (3 points), and language (9 points). The total score ranges from 0 to 30. A score of 24 or higher is considered indicative of normal cognitive function. The validity and reliability of the Turkish version of the test have been reported in the literature (r = 0.99)

CONTACTS AND LOCATIONS:
Overall Officials: Gulhan Yilmaz Gokmen, Assos. Prof., Study Chair — Bandırma Onyedi Eylül University
Locations (1):
- Bandirma Onyedi Eylul University, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No